CLINICAL TRIAL: NCT02953054
Title: A Double-Blind, Placebo-Controlled, Single-Dose Evaluation of the Dexmedetomidine Transdermal System for Post-Operative Analgesia Following Bunionectomy
Brief Title: Dexmedetomidine Transdermal System (DMTS) for Post-Operative Analgesia Following Bunionectomy
Acronym: DMTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPU-DMT-02-1503
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-06

CONDITIONS: Pain, Postoperative
Keywords: Pain; Bunionectomy; Dexmedetomidine; Transdermal; Patch; Postoperative; DMTS
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMTS (Active Comparator): DMTS applied to the upper arm
  Interventions: Drug: DMTS
- Placebo (Placebo Comparator): Placebo patches to match DMTS applied to the upper arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMTS — DMTS applied before surgery and worn for 72 hours
  Arms: DMTS
Drug: Placebo — Matching patches that have no active drug applied before surgery and worn for 72 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether the DMTS, compared with a placebo patch, will provide adequate pain relief during the first 3 days following bunionectomy surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the analgesic efficacy of the DMTS, compared with placebo in subjects with acute moderate to severe pain following unilateral bunionectomy.

The secondary objectives are:

* To assess the safety and tolerability of the DMTS, including assessment of skin irritation
* To assess adhesion of the DMTS
* To assess the sedation effect of the DMTS

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent.
2. Male or female, ≥ 18 years of age.
3. Scheduled to undergo a primary unilateral first metatarsal bunionectomy repair.
4. Have a physical status classification of 1 or 2 per the American Society of Anesthesiology.
5. Non-smoker for at least 1 year prior to screening; non-smoking is defined by cessation of smoking and use of all other tobacco and nicotine products (including chewing tobacco, snuff, e-cigarettes, nicotine patches, etc.).
6. Female subjects are eligible only if all the following apply:

   1. Not pregnant, not lactating, and not planning to become pregnant during the study
   2. Surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or have a same gender sex partner; or is practicing double-barrier contraception; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive
7. Male subjects with female sex partners must be surgically sterile or commit to the use of a reliable method of birth control.
8. Have a body weight > 50 kg, and body mass index of 22 to 38 kg/m2, inclusive.
9. Able to understand the study procedures, comply with all study procedures, and agree to participate in the study program for its full duration.

Exclusion Criteria:

1. Have a known sensitivity to dexmedetomidine or any excipient in the DMTS/placebo or to any peri- or postoperative medication whose use is required in this study.
2. Have a skin abnormality (eg, scar, tattoo) or unhealthy skin condition (eg, burns, wounds) at the patch application site, according to examination by the investigator at screening or admission to the clinic prior to surgery.
3. Have a clinically significant abnormal clinical laboratory test value.
4. Have history of or positive test results for the human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
5. Have a history or clinical manifestations of: a significant renal, hepatic, cardiovascular, metabolic, neurologic, or psychiatric condition; congestive heart failure, peptic ulcer, gastrointestinal bleeding, or other condition that would preclude participation in the study.
6. Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
7. Have another painful physical condition that may confound the assessments of postoperative pain.
8. Have a history of syncope or other syncopal attacks.
9. Have evidence of a clinically significant 12-lead ECG abnormality.
10. Have a history of alcohol abuse or prescription/illicit drug abuse.
11. Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol use at screening and/or clinic check-in.
12. Have a history or evidence of clinically significant orthostatic hypotension.
13. Have a resting heart rate of < 50 beats per minute or systolic blood pressure < 100 mmHg.
14. Have been receiving or have received opioid therapy chronically for > 2 weeks within the month prior to dosing of the study drug.
15. Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with dexmedetomidine.
16. Have had an upper respiratory tract infection within 14 days prior to dosing of the study drug.
17. Have utilized oral or injectable corticosteroids within 14 days prior to dosing of the study drug (intranasal and topical corticosteroid use during this time period is allowed).
18. Have received any investigational product within 30 days prior to dosing of the study drug.
19. Have previously received DMTS in a clinical trial.
20. Sensitivity to opioids, nonsteroidal anti-inflammatory drugs, or antibiotics.
21. In the opinion of the investigator or designee, is considered unsuitable for study entry and/or is unlikely to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-01-22 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Time-interval weighted summed pain intensity (SPI), measured using the 11 point (0 to 10) numeric rating scale (NRS) at designated time points from 4 to 24 hours following surgery (NRSSPI). | From 4 to 24 hours following surgery

SECONDARY OUTCOMES:
Time-interval weighted summed pain intensity over various time intervals | Up to 72 hours after surgery
The proportion of subjects using opioid rescue pain medication | Up to 72 hours after surgery
The time to first use of rescue pain medication | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: James Song, MS, MBA, Study Director — Teikoku Pharma USA, Inc.
Locations (2):
- Australia (2):
  - Nucleus Network LTD, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Background] Kivisto KT, Kallio A, Neuvonen PJ. Pharmacokinetics and pharmacodynamics of transdermal dexmedetomidine. Eur J Clin Pharmacol. 1994;46(4):345-9. doi: 10.1007/BF00194403. PMID 7957520
- [Background] Nemethy M, Paroli L, Williams-Russo PG, Blanck TJ. Assessing sedation with regional anesthesia: inter-rater agreement on a modified Wilson sedation scale. Anesth Analg. 2002 Mar;94(3):723-8; table of contents. doi: 10.1097/00000539-200203000-00045. PMID 11867405
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789